CLINICAL TRIAL: NCT02311166
Title: Soft Tissue Pathology in 100 Patients With Hip Dysplasia Before and After Periacetabular Osteotomy
Brief Title: Soft Tissue Pathology in Hip Dysplasia Before and After Periacetabular Osteotomy
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: 20140401PAO
Record Dates: First submitted 2014-04-02; First posted 2014-12-08 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2014-03

CONDITIONS: Hip Dysplasia
Keywords: Hip dysplasia; Soft tissue; Hip; Self-report; Physical activity
MeSH Terms: conditions — Hip Dislocation; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Introduction: The lack of congruence between the acetabulum and femoral head in hip dysplasia compromise the passive stability of the hip joint resulting in increased stress on the acetabular labrum, joint capsule and the muscles acting close to the hip joint. Soft tissue injury is present in hip dysplasia, and pathology of the iliopsoas muscle has been found in 18-50%. To our knowledge, no studies have systematically examined the prevalence of soft tissue pathology in hip dysplasia.

The overall aim of this research project is to examine soft tissue pathology in 100 patients with hip dysplasia prior to and one year after Periacetabular osteotomy (PAO).

Methods: Soft tissue pathology will be examined in a prospective cohort study on 100 patients with hip dysplasia prior to and one year after surgery. Pathology will be examined using ultrasonography and the Clinical Entities Approach that focus on pathology of the iliopsoas, adductors, rectus abdominis, gluteus medius and hamstrings. Furthermore, hip muscle strength is tested with a dynamometer, hip related health is measured with the Copenhagen Hip and Groin Outcome Score (HAGOS) and physical activity is measured with triaxial accelerometers during a period of 7 days.

Perspective: Is it possible to demonstrate pathology of the hip muscles and tendons applying clinical tests, muscle strength tests, and ultrasonography, as it has been found in sports-active people with groin pain, it will make sense to plan and test a specific training program focusing on the pathological soft tissue pathology.

DETAILED DESCRIPTION:
Introduction

In hip dysplasia the acetabulum presents as shallow and oblique with insufficient coverage of the femoral head. Deformity of the femoral neck and head is common with bilateral affection in 54%. The lack of congruence between the acetabulum and femoral head compromise the passive stability of the hip joint resulting in increased increased stress on the acetabular labrum, joint capsule and the muscles acting close to the hip joint. The increased stress on soft tissue results in acetabular labrum injury in 49-94% of the patients with hip dysplasia scheduled for joint preserving surgery. Left untreated hip dysplasia may lead to development of early osteoarthritis; however, the osteoarthritic process can be prevented or delayed with the Periacetabular osteotomy (PAO).

Soft tissue injury is present in hip dysplasia, and pathology of the iliopsoas muscle has been found in 18-50%. The muscles acting close to the hip joint including the deep fibers of the iliopsoas and the iliocapsularis muscle are together with the acetabular labrum and joint capsule able to increase the dynamic stabilisation of the femoral head in the dysplastic and shallow acetabulum. The hip joint is beside the iliopsoas further stabilised by the adductors and the gluteus medius muscle. Sustained hip pain and immobilisation has a negative impact on the iliopsoas, psoas and the hip adductors in terms of atrophy and decreased hip muscle strength. In an experimental study design it was found that decreased force contribution from the gluteal muscles during hip extension and the iliopsoas muscle during hip flexion resulted in an increase in the anterior hip joint force. The increased anterior hip joint force may contribute to anterior hip pain, subtle hip instability and the development of anterior acetabular labral tears.

Patients with hip dysplasia are less physical active prior to PAO mainly due to groin pain. A decreased physical activity level is likely to have a negative impact on the muscles acting close to the hip joint with a possible increased risk of sustaining further acetabular labrum injury and/or overuse related to soft tissue pathology. After surgery, the risk of overuse related soft tissue pathology might be further increased due to surgery impact on muscles and tendons. If it is possible to demonstrate pathology of the hip muscles and tendons applying clinical tests, muscle strength tests, and ultrasonography, as it has been found in sports-active people with groin pain, it will make sense to plan and test a specific training program focusing on the pathological soft tissue pathology.

The overall aim of this research project is to examine soft tissue pathology in 100 patients with hip dysplasia prior to and one year after PAO.

Material and methods

Design Prospective cohort study on 100 patients with symptomatic and radiologically verified hip dysplasia with one year of follow-up.

Inclusion

1. Diagnosis of hip dysplasia with a Wiberg´s Center-Edge (CE) angle <25 degrees, and planned PAO surgery at Aarhus University Hospital

Exclusion

1. Osteoarthritis grade ≥2 using Tönnis' classification
2. Other hip conditions as Calvé Perthes and epiphysiolysis
3. Surgery due to discus disease and spondylodesis and joint preserving and alloplastic surgery at the hip, knee or angle region
4. Neurological and/or rheumatological conditions affecting the function of the hip joint
5. Tenotomy of the iliopsoas tendon
6. BMI > 40
7. Cross-over sign (retroversion of the acetabulum)

Primary outcomes measures

1. Soft tissue pathology of abnormal clinical entities of the iliopsoas, adductors, rectus abdominis, gluteus medius and hamstrings using a standardized and reliable examination protocol
2. Soft tissue pathology of the iliopsoas, adductors, rectus abdominis, gluteus medius and hamstrings using a standardized ultrasonography protocol
3. Hip related health measured with the reliable Copenhagen Hip and Groin Outcome Score (HAGOS) validated on patients with groin pain
4. Physical activity measured with triaxial accelerometers during a period of 7 days on the following categories: rest, standing, walking, sit to stand (STS), cycling and running

Secondary outcome measures

1. Isometric hip muscle strength of the hip flexors, hip abductors, hip adductors and hip extensors using a reliable standardized method
2. Subjective visual analogue scale (VAS) at rest and during hip muscle strength tests
3. Pain location registered on a pain-drawing
4. Presence of internal snapping hip examined with a standardized examination test and ultrasonography
5. Presence of intra-articular pathology examined with the Flexion/Abduction/External Rotation (FABER) and Flexion/Adduction/Internal Rotation (FADDIR) tests and ultrasonography of the hip joint
6. Presence of lumbar and thoracic back pathology examined with the reliable Spine Springing Tests of the spinous process and processus transversi and of the sacrum
7. Conjoint tendon pathology examined with palpation of the pubic tubercle and ultrasonography of the pubic tubercle

Procedure

Patients are included from the division of hip surgery at Aarhus University Hospital using the listed inclusion and exclusion criteria's. The patients complete the HAGOS questionnaire after informed written consent. Wiberg's center-edge (CE) angle, Tönnis' acetabular index (AI) angle, and osteoarthritis grade are measured on anteroposterior radiographs after inclusion and after surgery by the surgeon. Information from the hospital charts is used to record age, gender, unilateral or bilateral involvement and other pathologies. Baseline characteristics are registered using standardized questions including data on BMI, duration of pain and intake of analgesia. Pain is afterwards measured on 100 mm visual analogue scale (VAS) resting in sitting and lying, and furthermore registered on a pain drawing. Preferred physical activity and hours spend on primary and overall physical activity is registered using standardized questions.

Ultrasonography is carried out first with an ultrasound scanner (Noblus, Hitachi-Aloka Medical, Zug, Switzerland) using an 18 Megahertz (MHz) linear transducer.Then the standardized examination protocol of abnormal clinical entities is carried out. Examination of pain at the conjoint tendon, presence of lumbar and thoracic back pathology, examination of intra-articular pathology and evaluation of internal snapping hip follow this. The hip muscle strength is then carried out, and finally the physical activity sensor is attached, and the patients are informed on how to monitor duration of physical activity.

One year postoperative the following examination is carried out in the listed order: HAGOS, baseline characteristics, pain on a VAS scale, pain on a pain drawing, hours of physical activity, ultrasonography, abnormal clinical entities, pain at the conjoint tendon, presence of lumbar and thoracic back pathology, examination of intra-articular pathology, evaluation of internal snapping hip, hip muscle strength. Finally the physical activity sensor is attached and the patient informed.

Statistics

Stata 11 is used for statistic calculations, and results are presented as significant if p<0.05.

Sample size

The present study is a descriptive study aiming to describe musculotendinous pathology in patients with hip dysplasia. This means that a power calculation is not feasible. On an annual basis approximately 140 periacetabular osteotomies is carried out on Aarhus University Hospital.

Allowing a lack of participation of 25 % it seems possible to include 100 patients during a period of one year. Based on this, a convenience sample of 100 patients is included to describe musculotendinous pathology in patients with hip dysplasia.

Ethics

The study was presented to the local research ethics the 14th of January 2014. The Committee waived the request of ethic approval, since the study according to Danish law does not require approval owing the observational design (Request 5/2014). All participants provided written consent prior to inclusion, and approval has been obtained from the Danish Data Protection Agency (Reference number: 1-16-02-47-14).

Economy and publicising

Financial support will be applied to internal and external funds. Both positive and negative results will be published in international journals and presented at conferences.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of hip dysplasia with a Wiberg´s Center-Edge (CE) angle <25 degrees, and planned PAO surgery at Aarhus University Hospital

Exclusion Criteria:

1. Osteoarthritis grade ≥2 using Tönnis' classification
2. Other hip conditions as Calvé Perthes and epiphysiolysis
3. Surgery due to discus disease and spondylodesis and joint preserving and alloplastic surgery at the hip, knee or angle region
4. Neurological and/or rheumatological conditions affecting the function of the hip joint
5. Tenotomy of the iliopsoas tendon
6. BMI > 40
7. Cross-over sign (retroversion of the acetabulum)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of hip dysplasia receiving treatment at Aarhus University Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Soft tissue pathology in the hip region (xamined with the Clinical Entities Approach) | Prior to surgery and one year after surgery
  Soft tissue pathology will be examined with the Clinical Entities Approach examining pathology of the iliopsoas, adductors, rectus abdominis, gluteus medius and hamstrings using a standardized and reliable examination protocol
Soft tissue pathology of the hip region using a standardized ultrasonography protocol | Prior to surgery and one year after surgery
  Soft tissue pathology of the iliopsoas, adductors, rectus abdominis, gluteus medius and hamstrings is examined using a standardized ultrasonography protocol.
Hip related self-reports of health (Copenhagen Hip and Groin Outcome Score (HAGOS) | Prior to surgery and one year after surgery
  Hip related health measured with the reliable Copenhagen Hip and Groin Outcome Score (HAGOS) validated on patients with groin pain.
Physical activity during a period of 7 days (measured with triaxial accelerometers) | Prior to surgery and one year after surgery
  Physical activity is measured with triaxial accelerometers during a period of 7 days on the following categories: rest, standing, walking, sit to stand (STS), cycling and running.

SECONDARY OUTCOMES:
Isometric hip muscle strength using a dynamometer | Prior to surgery and one year after surgery
  Isometric hip muscle strength of the hip flexors, hip abductors, hip adductors and hip extensors using a dynamometer
Subjective visual analogue scale (VAS) | Prior to surgery and one year after surgery
  Subjective visual analogue scale (VAS) at rest and during hip muscle strength tests.
Pain location registered on a pain-drawing | Prior to surgery and one year after surgery
  In an anatomical picture of a human body the patients records pain areas on the drawing.
Presence of internal snapping hip (examined with a standardized examination test) | Prior to surgery and one year after surgery
  Presence of internal snapping hip examined with a standardized examination test.
Presence of lumbar and thoracic back pathology | Prior to surgery and one year after surgery
  Presence of lumbar and thoracic back pathology is examined with the reliable Spine Springing Tests of the spinous process and processus transversi and of the sacrum.
Conjoint tendon pathology | Prior to surgery and one year after surgery
  Conjoint tendon pathology is examined with palpation of the pubic tubercle and ultrasonography of the pubic tubercle.

OTHER OUTCOMES:
Wiberg's center-edge (CE) angle | Prior to surgery and one year after surgery
  CE angel is measured on anteroposterior radiographs
Tönnis' acetabular index (AI) angle | Prior to surgery and one year after surgery
  Measured on anteroposterior radiographs
Osteoarthritis grade | Prior to surgery
  Measured on anteroposterior radiographs
Duration of pain | Prior to surgery
Intake of analgesia | Prior to surgery and one year after surgery
Preferred physical activity and hours spend on this | Prior to surgery and one year after surgery
Body Mass Index | Prior to surgery and one year after surgery
Age | Prior to surgery
Hours spend on general physical activity | Prior to surgery and one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, Prof. Dr.med, Study Chair — Department of Orthopaedic surgery, Aarhus University Hospital; Per Hölmich, Dr.med, Study Chair — Arthroscopic Center Amager, Amager University Hospital; Kristian Thorborg, MSc, PhD, Study Chair — Arthroscopic Center Amager, Amager University Hospital; Lars Bolvig, MD, Study Chair — Department of Orthopaedic surgery, Aarhus University Hospital; Stig S Jakobsen, MD, Study Chair — Department of Orthopaedic surgery, Aarhus University Hospital; Inger Mechlenburg, MSc, PhD, Study Director — Department of Orthopaedic surgery, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Orthopaedics, Aarhus University Hospital, Aarhus
  - Department of Physiotherapy and Occupational Therapy, Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: Undecided